CLINICAL TRIAL: NCT01796873
Title: Clopidogrel Resistance and Platelet Reactivity in Hispanic Females Undergoing Percutaneous Coronary Intervention
Brief Title: Clopidogrel Resistance and Platelet Reactivity in Women Undergoing Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0021-01
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2013-07

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Female; Hispanic; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Plavix (clopidogrel) is a drug that is approved by the FDA (Food and Drug Administration) to reduce the risk of having another heart attack by preventing platelets (blood cells that are important in forming blood clots) from sticking together and forming another clot. Platelet activity can be measured by a machine called VerifyNow.

The purpose of this study is to see whether Hispanic women and White non-Hispanic women have the same platelet response to a commonly used drug, Plavix (clopidogrel). Recent studies have shown that platelets may be more active in Hispanics, making it more difficult to prevent clots from forming, even when using Plavix. In addition, studies have shown that women may also have more active platelets than men. There have been no studies of Hispanic women and the effect of Plavix on platelet activity.

ELIGIBILITY:
Inclusion Criteria:

* All females age 45 or greater, presenting to University of Arizona Medical Center South Campus or University Campus Cardiology service with a history of ACS
* Hispanics will be defined via self-reporting as having both parents of Latino descent
* Currently taking clopidogrel

Exclusion Criteria:

* Taking any of the following antiplatelet drugs:

  * Prasugrel (Effient)
  * Ticagrelor (Brilinta)
  * Ticlopidine (Ticlid)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females, age ≥ 45 years, with Acute Coronary Syndrome (ACS), undergone a percutaneous coronary intervention and currently treated with clopidogrel will be enrolled. The subjects' race and ethnicity will be self -reported and Hispanic ethnicity by self-report of having both parents of Hispanic/Latino descent.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity measured by the VerifyNow P2Y12 Assay | At least 14 days following the ACS event
  Compare the Hispanic female platelet reactivity response to the Caucasian female platelet reactivity response in females currently taking clopidogrel.

CONTACTS AND LOCATIONS:
Overall Officials: Sasanka Jayasuriya, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona Medical Center South Campus, Tucson, Arizona
  - University of Arizona Medical Center University Campus, Tucson, Arizona

REFERENCES:
- [Background] Frelinger AL 3rd, Bhatt DL, Lee RD, Mulford DJ, Wu J, Nudurupati S, Nigam A, Lampa M, Brooks JK, Barnard MR, Michelson AD. Clopidogrel pharmacokinetics and pharmacodynamics vary widely despite exclusion or control of polymorphisms (CYP2C19, ABCB1, PON1), noncompliance, diet, smoking, co-medications (including proton pump inhibitors), and pre-existent variability in platelet function. J Am Coll Cardiol. 2013 Feb 26;61(8):872-9. doi: 10.1016/j.jacc.2012.11.040. Epub 2013 Jan 16. PMID 23333143
- [Background] Wenaweser P, Daemen J, Zwahlen M, van Domburg R, Juni P, Vaina S, Hellige G, Tsuchida K, Morger C, Boersma E, Kukreja N, Meier B, Serruys PW, Windecker S. Incidence and correlates of drug-eluting stent thrombosis in routine clinical practice. 4-year results from a large 2-institutional cohort study. J Am Coll Cardiol. 2008 Sep 30;52(14):1134-40. doi: 10.1016/j.jacc.2008.07.006. PMID 18804739
- [Background] Baber U. et al., Impact of Self-Reported Ethnicity on Response to Clopidogrel in Patients Undergoing Percutaneous Coronary Intervention. Circulation. 2010;122:A20850